CLINICAL TRIAL: NCT06497101
Title: Effectiveness of Temperament Based Therapy With Support (TBT-S): A Novel 5-day Treatment for Anorexia Nervosa
Brief Title: Effectiveness Trial of Temperament Based Therapy With Support (TBT-S)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Kristin Stedal, Senior Researcher, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 728279
Record Dates: First submitted 2024-07-04; First posted 2024-07-11 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Temperament Based Therapy with Support (TBT-S) (Experimental): TBT-S in addition to treatment as usual
  Interventions: Behavioral: Temperament Based Therapy with Support (TBT-S)
- Treatment as Usual (TAU) (No Intervention): Treatment as Usual

INTERVENTIONS:
Behavioral: Temperament Based Therapy with Support (TBT-S) — Participants included in the intervention arm will receive TBT-S (5-day treatment) in addition to treatment as usual (TAU)
  Other Names: TBT-S
  Arms: Temperament Based Therapy with Support (TBT-S)

SUMMARY:
The main aim of this project is to determine the short and long-term effectiveness of an out-patient treatment for patients with anorexia nervosa. Specifically, we will measure whether TBT-S in addition to treatment as usual (TAU) will be more effective than TAU alone in reducing eating disorder psychopathology. Assessments will be conducted at four timepoints; pre and post TBT-S, and at 3 and 12 months follow-up. Primary outcome measure is eating disorder psychopathology, with the hypothesis that patients receiving TBT-S in addition to TAU will show significantly greater reduction in eating disorder psychopathology from TBT-S treatment admission to 3 month follow-up, compared to controls.

DETAILED DESCRIPTION:
Participants in the intervention arm will receive five days of TBT-S in addition to treatment as usual. TBT-S is administered to three to six adult anorexia nervosa patients with up to four supports per patient. The treatment structure consists of five consecutive days of treatment, up to 7,5 hours each day. Staff requirements for TBT-S are three clinicians, one dietician and one medical staff. Adults referred to a local psychiatric centre (DPS) for out-patient anorexia nervosa treatment, and their supports, will be eligible to participate in the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18, all genders
* A Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnosed anorexia nervosa disorder (F50.0, F50.01, F50.02, also including F50.9 - atypical anorexia nervosa)
* Willingness to have Support(s) participate in treatment
* Medically stable

Exclusion Criteria:

* Diagnosis of Intellectual Disability or Schizophrenia spectrum/other psychotic disorder
* Diagnosis of alcohol or drug abuse or dependence in the 3 months prior to the study
* Receiving in-patient treatment at time of study entry
* Presence of other psychopathology that might interfere with ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Psychopathology | Baseline, after 1 week and at 3 and 12 months follow-up
  Eating Disorders Examination Questionnaire (EDE-Q). Participants report symptomatology on a 7-point Likert scale from 0 (no days) to 6 (everyday). The EDE-Q contains 4 subscales: Restraint, Weight Concern, Eating Concern, and Shape Concern. Subscale scores are calculated by finding the averages of the subscale items. A global score is also calculated by averaging the subscale scores. Scores range from 0 to 6; higher scores indicate higher levels of eating disorder pathology.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Regional Department for Eating Disorders, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No
There are no plans to make individual participant data (IPD) available to other researchers.